CLINICAL TRIAL: NCT07278947
Title: Effects of an Online Psychoeducational and Psychotherapeutic Programme for Caregivers of Children With Hearing Loss Post-Cochlear Implantation: A Pilot Randomised Controlled Trial
Brief Title: ACT-based Parenting Program for Caregivers of Children With Hearing Loss Post-cochlear: A Pilot Randomised Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: Xiangya Hospital of Central South University (Other); The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Jiao Xie, Associate Chief Nurse, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: LYEC2025-0209
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Hearing Loss; Stress; Depression, Anxiety
MeSH Terms: conditions — Hearing Loss; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Two arm, pretest posttest, assessor blinded Randomised Controlled Trial (RCT)
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Eligible parents consenting to participate will be randomly assigned to either the Intervention (ACT-based parenting program) or Control (usual-care) Group in a 1:1 ratio, using the permuted block size of 4 through sequentially numbered, opaque and sealed envelopes with number cards (1=intervention, 2=control). A separate set of random numbers, concealed from the research team and RAs, will be generated by a statistician. Clerical staff uninvolved in the project will administer the randomisation. The research assistant (RA-1), blinded to subject selection, will open the envelopes only after informed consent and baseline assessments are completed. The research assistant (RA-2) is also blinded to group assignments and will conduct assessments/evaluations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT-based parenting program+usual care (Experimental): Parents will receive 6 ACT-based parenting program sessions, one weekly session, 45-60 mins per session. These sessions will be one-on-one, conducted via video conferencing.
  Interventions: Behavioral: ACT-based parenting program+usual care
- Usual care (Active Comparator): Parents will receive usual care delivered by otology nurses regarding post-cochlear implantation care instructions.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: ACT-based parenting program+usual care — The ACT-based parenting program integrates two complementary components: (1) targeted psychoeducation on post-CI care (device use and troubleshooting, home-based auditory rehabilitation, realistic progress monitoring, school and social participation, communication strategies, and navigation of rehabilitation services); and (2) brief, skills-focused psychotherapeutic content grounded in ACT principles to enhance psychological flexibility (e.g., present-moment awareness, defusion from difficult thoughts, acceptance of difficult emotions and sensations, values clarification, and committed action in daily caregiving). By combining condition-specific knowledge with process-based skills, the intervention is designed to address both informational needs and core psychopathological processes that perpetuate caregiver distress.
  Arms: ACT-based parenting program+usual care
Other: Usual care — Parents in the control arm will receive usual care delivered by otology nurses covering post-cochlear implantation care instructions (e.g., device safety, basic troubleshooting, follow-up schedules) and will have access to standard rehabilitation services as per clinic routines. After final assessments, waitlist participants may be offered access to intervention materials where appropriate.
  Arms: Usual care

SUMMARY:
The purpose of the proposed pilot randomized controlled design study is to evaluate the feasibility, acceptability, and potential effectiveness of using a videoconferencing-based individual Acceptance and Commitment Therapy (ACT) approach to enhance the mental well-being and parenting competence of parents of children with hearing loss post-cochlear implantation over a three-month period after the intervention has taken place.

DETAILED DESCRIPTION:
Caregivers of children with hearing loss post-cochlear implantation (CI), experience sustained caregiving demands that place them at elevated risk for stress, anxiety, depressive symptoms, and reduced family functioning. The postoperative journey commonly involves intensive device mapping, auditory-verbal therapy, daily home-based training, and frequent medical or rehabilitation appointments. These demands, coupled with uncertainty about the child's auditory, speech, and psychosocial outcomes, can erode caregiver well-being and strain family routines. Evidence across populations indicates that psychoeducational and psychotherapeutic interventions can improve caregiver mental health and parenting efficacy by providing knowledge, skills, and strategies that enhance coping and resilience.

Acceptance and Commitment Therapy (ACT) and related third-wave approaches have shown benefits for parents of children with chronic conditions by increasing psychological flexibility-an empirically supported process linked to improved mental health and adaptive caregiving. However, prior trials in similar caregiver populations have sometimes yielded modest effect sizes, in part due to high resource requirements (e.g., reliance on extensively trained therapists) and insufficient focus on the most impaired transdiagnostic processes (e.g., cognitive fusion, experiential avoidance, values-behavior disconnect). In addition, access barriers (time, travel, childcare) limit uptake of in-person programs, especially for families navigating intensive post CI rehabilitation schedules.

This pilot randomized controlled trial (RCT) will evaluate the feasibility, acceptability, and preliminary effectiveness of an online psychoeducational and psychotherapeutic programme tailored for caregivers of children with hearing loss following cochlear implantation. The programme integrates two complementary components: (1) targeted psychoeducation on post CI care (device use and troubleshooting, auditory rehabilitation at home, realistic progress monitoring, school and social participation, communication strategies, and navigation of rehabilitation services); and (2) brief, skills focused psychotherapeutic content grounded in ACT principles to enhance psychological flexibility (e.g., present moment awareness, defusion from difficult thoughts, acceptance of difficult emotions and sensations, values clarification, and committed action in daily caregiving). By combining condition specific knowledge with process based skills, the intervention is designed to address both informational needs and core psychopathological processes that perpetuate caregiver distress.

The programme will be delivered via secure videoconferencing in a structured, time limited format to reduce burden and improve accessibility. Sessions will include didactic micro modules, guided experiential exercises (e.g., mindfulness, values mapping, defusion techniques), and applied practice tied to real world caregiving tasks (e.g., integrating values into daily listening practice, using brief acceptance/defusion skills during child resistance to wear time, and problem solving around school or therapy transitions). Between-session activities will reinforce learning through short videos, worksheets, and practice logs. Content will be developmentally and culturally adapted for families of children using CIs, with attention to diverse communication modalities and family preferences.

Participants will be randomly assigned to the online programme or a waitlist control. Outcome assessments will occur at baseline (pre intervention) and immediately post intervention. Primary feasibility and acceptability metrics will include recruitment, retention, session attendance, completion of between session activities, and participant-rated satisfaction and perceived usefulness. Preliminary effectiveness outcomes will focus on caregiver mental health and functioning (e.g., stress, anxiety/depressive symptoms, psychological flexibility, and parenting self efficacy). Exploratory outcomes will include family functioning, adherence to home auditory verbal practice, and caregiver reported child participation in everyday listening and communication activities.

We hypothesize that the online programme will be feasible and acceptable to caregivers and will yield greater improvements than usual-care-only control in caregiver mental health, psychological flexibility, and parenting self-efficacy from baseline to post intervention. By using a brief, process based approach and remote delivery, the intervention aims to lessen reliance on scarce specialist time, reduce participation barriers, and target the mechanisms most closely linked to caregiver distress. Findings from this pilot will inform refinement of content, dosing, and implementation strategies, and will provide effect size estimates to power a future full scale RCT.

ELIGIBILITY:
Inclusion Criteria:

1. Mandarin-speaking Chinese residents aged ≥18 years.
2. Their child is scheduled to undergo cochlear implant surgery within the next month or has undergone cochlear implant surgery within the past month.
3. Living with their child with hearing loss who uses (or will use) a cochlear implant.
4. Primary caregiver responsible for the child's daily care.
5. Has reliable internet access via a computer and/or smartphone for video-conferencing (e.g., TenCent Meeting, Zoom) and is willing to maintain access for the duration of the intervention.

Exclusion Criteria:

1. Parents with cognitive deficiency, severe mental illness and/or disability conditions that interfere with their ability to comprehend the programme's content.
2. Current substance or alcohol dependence.
3. Pregnancy or postpartum period (<6 months).
4. Participation in any ACT-based intervention within the past six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Parental Stress | Change from baseline assessment to immediate post-intervention
  The Parental Stress Scale (PSS, 18-item, 5-point scale) will assess parenting stress. A higher score represents a higher level of parental stress. The Chinese version of the PSS has demonstrated acceptable psychometric properties and is therefore suitable for use by researchers to assess the parental stress levels of Chinese parents.

SECONDARY OUTCOMES:
Parental depressive symptoms | Change from baseline assessment to immediate post-intervention
  The Patient Health Questionnaire (PHQ-9, 9-item, 4-point Likert scale) will be used to assess the frequency of the parents experiencing depressive symptoms in the past two weeks. The Chinese version of the PHQ-9 has demonstrated good internal consistency reliability (Cronbach's alpha = 0.86) and test-retest correlation coefficient.
Parental anxiety symptoms | Change from baseline assessment to immediate post-intervention
  The Generalized Anxiety Disorder-7 (GAD-7, 7-item, 4-point Likert scale) will be used to measure the severity of anxiety symptoms. The Chinese version of the GAD-7 demonstrated good reliability and validity with a Cronbach's coefficient of 0.91.
Parental Psychological Flexibility | Change from baseline assessment to immediate post-intervention
  The PsyFlex (5-point Likert scale, 6 items) will be used to assess the six therapeutic processes in ACT, namely contacting the present moment, defusion, acceptance, self-as-context, values and committed action.
Parenting competency | Change from baseline assessment to immediate post-intervention
  The Parenting Sense of Competence Scale (PSOC, 17-item, 6-point Likert scale) will be used to measure the level of parenting competency. The Chinese version of the PSOC demonstrate good reliability and validity with a Cronbach's coefficient of 0.87.
Satisfaction of the intervention | This outcome will be assessed 1-2 weeks after the end of the intervention.
  The 18-item self-developed intervention satisfaction questionnaire and a group qualitative interview will be conducted 1-2 weeks after the end of the intervention. The satisfaction form, adopted from the 15-item self-reported Chinese Standardized Client Satisfaction Scale (C-SCS), utilized a 5-point Likert-scale to measure satisfaction with intervention design, duration, components, intervener performance, accessibility, needs fulfillment, and overall satisfaction.

IPD SHARING:
Plan to Share IPD: No
Considering ethical reasons and participant privacy, we will not make individual participant data publicly available.